CLINICAL TRIAL: NCT01360554
Title: Archer 1009:a Randomized, Double Blind Phase 3 Efficacy And Safety Study Of Pf-00299804 (Dacomitinib) Versus Erlotinib For The Treatment Of Advanced Non-small Cell Lung Cancer Following Progression After, Or Intolerance To, At Least One Prior Chemotherapy
Brief Title: ARCHER 1009 : A Study Of Dacomitinib (PF-00299804) Vs. Erlotinib In The Treatment Of Advanced Non-Small Cell Lung Cancer
Acronym: ARCHER 1009
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A7471009; 2010-022656-22 (EudraCT Number)
Record Dates: First submitted 2011-04-12; First posted 2011-05-25 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: comparative study of PF-00299804 and Erlotinib; Double-Blind Phase 3 trial of TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Blinded active PF-00299804 + blinded placebo comparator (erlotinib)
  Interventions: Drug: Dacomitinib (PF-00299804); Drug: Placebo erlotinib
- B (Active Comparator): Blinded active comparator (erlotinib) + blinded placebo PF-00299804
  Interventions: Drug: Active Comparator (erlotinib); Drug: Placebo PF00299804

INTERVENTIONS:
Drug: Dacomitinib (PF-00299804) — Dacomitinib (PF-00299804) is provided as 45 mg tablets, continuous oral daily dosing
  Arms: A
Drug: Active Comparator (erlotinib) — Active comparator (erlotinib) provided as 150 mg tablet, continuous oral daily dosing
  Arms: B
Drug: Placebo erlotinib — placebo erlotinib, provided as 150 mg tablet, continuous oral daily dosing.
  Arms: A
Drug: Placebo PF00299804 — placebo PF-00299804, provide as 45 mg tablet, continuous oral daily dosing
  Arms: B

SUMMARY:
This is a multinational, multicenter, randomized,double-blinded, Phase 3 study comparing the efficacy and safety of treatment with PF-00299804 to treatment with erlotinib in patients with advanced non-small cell lung cancer, previously treated with at least one prior regimen. Analyses of primary objective (Progression Free Survival) will be done in two co-primary populations as defined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of pathologically confirmed, advanced NSCLC (with known histology).
* Prior treatment with at least one and no more than two systemic therapy regimens (at least one must be standard chemotherapy for advanced NSCLC).
* Adequate tissue sample must be submitted prior to randomization for tumor biomarker analyses.
* Adequate renal, hematologic, liver function.
* ECOG PS of 0-2.
* Radiologically measurable disease.

Exclusion Criteria:

* Small cell histology.
* Symptomatic brain mets or known leptomeningeal mets.
* Prior therapy with agent known or proposed to be active by action on EGFR tyrosine kinase or other HER family proteins.
* Uncontrolled medical disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2011-06-16; Primary Completion 2013-09-30 (Actual); Study Completion 2015-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (221):
- United States (105):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwest Alabama Cancer Center, Florence, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Ironwood physicians P C dba Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Chandler, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Gilbert, Arizona
  - Desert Oncology Associates dba Ironwood Cancer and Research Centers, Mesa, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer and Research Centers, Mesa, Arizona
  - Highlands Oncology Group PA, Fayetteville, Arkansas
  - Highlands Oncology Group, PA, Rogers, Arkansas
  - Central Hematology Oncology Medical Group Inc., Alhambra, California
  - UCLA Hematology Oncology-Alhambra, Alhambra, California
  - City of Hope, Duarte, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Drug Management Only, Los Angeles, California
  - Drug Managerrent Only:, Los Angeles, California
  - UCLA West Medical Pharmacy, Los Angeles, California
  - Administrative Address: UCLA Hematology Oncology-Clinical Research Unit (CRU), Los Angeles, California
  - Drug Shipment Address: Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - Regulatory Management Only:, Los Angeles, California
  - Regulatory Management:, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - TORI Central Administration, Los Angeles, California
  - Westwood Bowyer Clinic, Peter Morton Medical Building, Los Angeles, California
  - UCLA/Pasadena Healthcare Hematology-Oncology, Pasadena, California
  - Central Hematology Oncology Medical Group, Inc., Pasadena, California
  - Cancer Care Associates Medical Group Inc., Redondo Beach, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Hematology Oncology-Parkside, Santa Monica, California
  - UCLA Hematology Oncology-Santa Monica, Santa Monica, California
  - UCLA Santa Monica Medical Center & Orthopedic Hospital, Santa Monica, California
  - City of Hope South Pasadena Cancer Center, South Pasadena, California
  - UCLA/Santa Clarita Valley Cancer Center, Valencia, California
  - UCLA Cancer Center, Westlake Village, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Florida Hospital, Orlando, Florida
  - Cancer Institute of Florida, Orlando, Florida
  - Hematology and Oncology Consultants, P.A., Orlando, Florida
  - Investigational Drug Services, Florida Hospital, Orlando, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, P.C., Austell, Georgia
  - Northwest Georgia Oncology Centers, P.C., Carrollton, Georgia
  - Northwest Georgia Oncology Centers, PC, Cartersville, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Atlanta Cancer Care, Decatur, Georgia
  - Georgia Cancer Specialists, Decatur, Georgia
  - The Cancer Center at DeKalb Medical, Decatur, Georgia
  - Northwest Georgia Oncology Centers, P.C., Douglasville, Georgia
  - Suburban Hematology-Oncology Associates, P.C., Duluth, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oncology Specialists of North Georgia, LLC, Gainesville, Georgia
  - The Longstreet Clinic Cancer Center, Gainesville, Georgia
  - Suburban Hematology-Oncology Associates, P.C., Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Suburban Hematology-Oncology Associates, P.C., Snellville, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Ingalls Memorial Hospital - In-Patient Pharmacy, Harvey, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Monroe Medical Associates, Harvey, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Monroe Medical Associates, Tinley Park, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Cedar Valley Medical Specialists, P.C., Waterloo, Iowa
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - University Medical Center, Inc., Louisville, Kentucky
  - University Medical Center, Inc, Louisville, Kentucky
  - Baptist Hospital East, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at Farmington Hills, Farmington Hills, Michigan
  - North Mississippi Hematology and Oncology Associates, Ltd., Starkville, Mississippi
  - North Mississippi Hematology and Oncology Associates, Ltd.,, Tupelo, Mississippi
  - Siteman Cancer Center-St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center-West County, Creve Coeur, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine-IDS Pharmacy, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center /Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Oncology and Hematology Specialists, P.A., Denville, New Jersey
  - Stony Brook University-Cancer Center, Stony Brook, New York
  - Carolina Oncology Specialists PA, Hickory, North Carolina
  - Carolina Oncology Specialists PA, Lenoir, North Carolina
  - Mercy clinic oklahoma communities, Inc. - Mercy clinic oncology/Hematology - Norman, Norman, Oklahoma
  - Mercy Physicians of Oklahoma-Communities, Inc. - Mercy Clinic Oncology/Hematology - McAuley, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City - Oncology Infusion, Oklahoma City, Oklahoma
  - Good Samaritan Hospital Samaritan Ambulatory Infusion Services, Corvallis, Oregon
  - Samaritan Hematology & Oncology Consultants, Corvallis, Oregon
  - Samaritan Pharmacy Services, Corvallis, Oregon
  - Samaritan North Lincoln Hospital, Lincoln City, Oregon
  - Samaritan Pacific Communities Hospital, Newport, Oregon
  - Guthrie Clinic, Limited, Sayre, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Kadlec Medical Center, Richland, Washington
  - Outpatient Imaging Center, Richland, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Sozialmedizinisches Zentrum Baumgartner Hoehe - Otto Wagner Spital und Pflegezentrum, Vienna, Austria
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Laboratoire de la Porte de Hall, Brussels
  - Grand Hopital de Charleroi Oncologie-Hematologie, Charleroi
  - CHU Ambroise Parre- Service Biologie Clinique, Mons
  - Heilig Hart Ziekenhuis Roeselare-Menen, Roeselare
- China (5):
  - Tumour Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology/Cancer Center, Wuhan, Hubei
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Shanghai Pulmonary Hospital, Shanghai
- Aalborg Sygehus Syd, Aalborg, Denmark
- Finland (2):
  - Helsingin yliopistollinen sairaala, Meilahden kolmiosairaala, keuhkosairauksien poliklinikka, Helsinki
  - Satakunnan keskussairaala/Keuhkosairauksien osasto A4, Pori
- France (5):
  - Centre Georges Francois Leclerc, Dijon
  - Hopital Albert Michallon, Grenoble
  - Hôpital Paris Saint Joseph, Paris
  - CHU de Poitiers, Poitiers
  - Institut de Cancerologie de lOuest - Rene Gauducheau, Saint-Herblain
- Germany (5):
  - Universitaetsklinikum Aachen, Aachen
  - Asklepios Fachkliniken Muenchen-Gauting, Gauting
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet, Mainz
  - Krankenhaus Bethanien, Medizinische Klinik III, Moers
- Greece (3):
  - University Hospital of Larissa, Larissa, Thessaly
  - Sotiria General Hospital of Athens, Athens
  - University Hospital of Heraklion, Heraklion
- Hungary (6):
  - Semmelweis Egyetem Pulmonologiai Klinika, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Veszprem Megyei Onkormanyzat Tudogyogyintezete, Farkasgyepű
  - Pandy Kalman Megyei Korhaz, Aktiv Tudogyogyaszat, Gyula
  - Josa Andras Oktatokorhaz Egeszsegugyi Szolgaltato Nonprofit Kft., Nyíregyháza
  - Zala Megyei Korhaz, Pulmonologiai Osztaly, Zalaegerszeg-Pozva
- India (4):
  - Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Manipal Hospital, Bangalore, Karnataka
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
- Ireland (4):
  - St Vincent's University Hospital, Dublin, Leinster
  - Beaumont Hospital, Dublin, Leinster
  - St. James Hospital, Dublin
  - Oncology Department, Waterford
- Japan (20):
  - Aichi cancer center central hospital /Thoracic Oncology, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City General Hospital Department of Clinical Oncology, Osaka, Osaka
  - Kinki University Hospital, Osakasayama-shi, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai-Shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - National Hospital Organization, Yamaguchi-Ube Medical Center, Ube-shi, Yamaguchi
  - National Hp. Org. Kyushu Medical Center, Fukuoka
  - National Hospital Organization Kyushu Cancer Center/Department of Thoracic Oncology, Fukuoka
  - Kyushu University Hospital Respiratory Medicine, Fukuoka
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- Oaxaca Site Management Organization, Oaxaca City, Mexico
- Poland (4):
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock, Masovian Voivodeship
  - Zoz All-Medi, Otwock, Masovian Voivodeship
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Nukleomed, Warsaw, Masovian Voivodeship
- Russia (11):
  - City Hospital #2 Krasnodar Multi-Field Diagnostic and Treatment Association, Krasnodar, Krasnodarskiy Kray
  - Oncology Center # 2, Sochi, Krasnodarskiy Kray
  - Federal State Healthcare Clinical Hospital #101 of the Federal Biomedical Agency, Pyatigorsk, Stavropolskij Kraj
  - Pyatigorsk Oncology Center, Pyatigorsk
  - Clinic of Hospital Surgery, Saint Petersburg
  - Military Medical Academy n.a. S.M.Kirov, Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - St.-Petersburg State Medical University I.P.Pavlov of Roszdrav, Saint Petersburg
  - Research Institute of Pulmonology, Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg
  - Samara Regional Clinical Oncology Dispensary, Samara
- Slovakia (3):
  - Univerzitna Nemocnica Bratislava, Klinika pneumologie a ftizeologie I- Oddelenie klinickej onkologie, Bratislava
  - Specializovana nemocnica sv. Svorada Zobor, n.o., Nitra
  - Fakultna nemocnica s poliklinikou, Nové Zámky
- South Africa (4):
  - WCR: Wits Clinical Research, Parktown,Johannesburg, Gauteng
  - GVI Oncology Clinical Research Unit, Kraaifontein, Western Cape
  - Department of Oncotherapy, Bloemfontein
  - GVI Oncology, Port Elizabeth
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Clinical Trial Center, Seoul
  - Asan Medical Center, Department of Oncology, Seoul
- Spain (14):
  - Hospital General Universitario de Elche - Edificio UIAE, Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Provincial de Castellon - Servicio de Oncologia, Castellon, Castellon
  - HOSPITAL DE LA SANTA CREU I SANT PAU - Pharmacy, Barcelona
  - Hospital de la Santa Creu i Sant Pau - AGDAC, Barcelona
  - Hospital de la Santa Creu i Sant Pau - Anatomia Patológica, Barcelona
  - Hospital de la Santa Creu i Sant Pau - Diagnostic per la Imatge i Med. Nuclear, Barcelona
  - Hospital de la Santa Creu i Sant Pau - Hospital de Día, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Provincial de Castellon (Farmacia), Castellon
  - Hospital Universitario 12 de Octubre-Radiology, Madrid
  - Hospital Universitario 12 de Octubre01, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio. Hospital General Planta Baja. Servicio de Oncologia., Seville
- Sweden (2):
  - KPE/Onkologikliniken, Karlstad
  - Karolinska Universitetssjukhuset, Stockholm
- Switzerland (5):
  - Kantonsspital Aarau, Aarau
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Hopitaux Universitaires de Geneve, Geneva
  - Ospedale Regionale di Locarno La Carita, Locarno
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (8):
  - Kent Oncology Centre, Maidstone, Kent
  - New Cross Hospital - Royal Wolverhampton Hospital NHS Trust, Wolverhampton, West Midlands
  - North Middlesex NHS Trust, Edmonton
  - Leicester Royal Infirmary, Leicester
  - Cancer Clinical Trials Unit, London
  - Christie Hospital NHS Trust, Department of Medical Oncology, Manchester
  - Christie Hospital NHS Trust, Manchester
  - Lung and Melanoma Research Team, Manchester

REFERENCES:
- [Derived] Ramalingam SS, O'Byrne K, Boyer M, Mok T, Janne PA, Zhang H, Liang J, Taylor I, Sbar EI, Paz-Ares L. Dacomitinib versus erlotinib in patients with EGFR-mutated advanced nonsmall-cell lung cancer (NSCLC): pooled subset analyses from two randomized trials. Ann Oncol. 2016 Mar;27(3):423-9. doi: 10.1093/annonc/mdv593. Epub 2016 Jan 13. PMID 26768165
- [Derived] Ramalingam SS, Janne PA, Mok T, O'Byrne K, Boyer MJ, Von Pawel J, Pluzanski A, Shtivelband M, Docampo LI, Bennouna J, Zhang H, Liang JQ, Doherty JP, Taylor I, Mather CB, Goldberg Z, O'Connell J, Paz-Ares L. Dacomitinib versus erlotinib in patients with advanced-stage, previously treated non-small-cell lung cancer (ARCHER 1009): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1369-78. doi: 10.1016/S1470-2045(14)70452-8. Epub 2014 Oct 15. PMID 25439691
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471009&StudyName=ARCHER%201009%20%3A%20A%20Study%20Of%20Dacomitinib%20%28PF-00299804%29%20Vs.%20Erlotinib%20In%20The%20Treatment%20Of%20Advanced%20Non-Small%20Cell%20Lung%20Cancer%20%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 134 sites with 878 participants randomized in a 1:1 ratio to 1 of 2 treatment arms, of these 872 were treated. Eligible participants who provided written informed consent and met all inclusion and exclusion criteria were assigned a Single Subject Identification number and randomized by the central randomization system.
Pre-assignment Details: There were no significant study milestones following participant enrollment, but prior to group assignment.
Groups:
- Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo): Participants randomized to Arm A received dacomitinib 45 mg orally once daily and erlotinib 150 mg placebo orally once daily. Participants began treatment within 3 days after randomization and continued treatment without breaks until they experienced unacceptable toxicity, tumor progression, or death.
- Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo): Participants randomized to Arm B received erlotinib 150 mg orally once daily and dacomitinib 45 mg placebo orally once daily. Participants began treatment within 3 days after randomization and continued treatment without breaks until they experienced unacceptable toxicity, tumor progression, or death.
Period: Overall Study
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Started | 439 (Three participants were randomized but not treated.) | 439 (Three participants were randomized but not treated.)
Treated | 436 | 436
Completed | 0 | 0
Not Completed | 439 | 439
Not completed — Death | 359 | 371
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 23 | 24
Not completed — Study terminated by sponsor | 49 | 37
Not completed — Other, not specified | 1 | 0
Not completed — Randomized but not treated. | 3 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo) | Total
Number analyzed (Participants) | 436 | 436 | 872
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.57) | 61.7 (9.71) | 62.5 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 161 | 311
  Male | 286 | 275 | 561

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Independent Radiologic Review.
Description: PFS was defined as the time from randomization to the date of disease progression as by Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 per Independent Radiologic Review or death due to any cause, whichever occurred first. Objective progression was defined as a 20% increase in the sum of the diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions, or the appearance of any new unequivocal malignant lesions.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, participants were followed up until progressive disease regardless of start of subsequent cancer therapy.
Population: The ITT population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether patients received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 439 | 439
Months | 2.6 [1.9 to 2.8] | 2.5 [1.9 to 2.8]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Test type: Superiority or Other; p = 0.195, 1-sided stratified log-rank test — One-sided P-value; Stratified by epidermal growth factor receptor (EGFR) status, Kirsten Rat Sarcoma status (KRAS), baseline Eastern Cooperative Oncology Group (ECOG); Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.797 to 1.093] — The HR (Dacomitinib arm versus erlotinib arm) and 95% CI were estimated from stratified Cox regression with EGFR status, KRAS, baseline ECOG as stratification factors

2. Primary Outcome: Progression-Free Survival (PFS) Per Independent Radiologic Review in KRAS Wild-type (WT) Participants.
Description: PFS was defined as the time from randomization to the date of disease progression as by RECIST v1.1 per Independent Radiologic Review or death due to any cause, whichever occurred first. Objective progression was defined as a 20% increase in the sum of the diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions, or the appearance of any new unequivocal malignant lesions. Tumor tissue from participants' original diagnostic biopsies or recently obtained biopsies were analyzed to determine KRAS status.
Time Frame: as for outcome 1
Population: ITT population for KRAS-WT participants: all participants who were confirmed as having KRAS-WT tumors, randomized, with study drug assignment designated according to initial randomization, regardless of whether patients received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 256 | 263
Months | 2.6 [1.9 to 2.9] | 2.5 [1.9 to 3.0]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Test type: Superiority or Other; p = 0.643, 1-sided stratified log-rank test — One-sided P-value; Stratified by EGFR status and baseline ECOG; Hazard Ratio (HR) = 1.037, 95% CI 2-sided [0.848 to 1.268] — The HR (Dacomitinib arm versus erlotinib arm) and 95% CI were estimated from stratified Cox regression with EGFR status and baseline ECOG as stratification factors

3. Secondary Outcome: PFS Based on Investigator Review.
Description: PFS was defined as the time from randomization to the date of disease progression as by RECIST v1.1 per Investigator's Review or death due to any cause, whichever occurred first. Objective progression was defined as a 20% increase in the sum of the diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions, or the appearance of any new unequivocal malignant lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 439 | 439
Months | 1.9 [1.9 to 2.6] | 1.9 [1.8 to 2.1]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Test type: Superiority or Other; p = 0.069, 1-sided stratified log-rank test — Stratified by EGFR status, KRAS status, and baseline ECOG; One-sided P-value; Hazard Ratio (HR) = 0.899, 95% CI 2-sided [0.780 to 1.035] — The HR (Dacomitinib arm versus erlotinib arm) and 95% CI were estimated from stratified Cox regression with EGFR status, KRAS status, and baseline ECOG as stratification factors

4. Secondary Outcome: PFS Based on Investigator Review in KRAS-WT Participants.
Description: PFS was defined as the time from randomization to the date of disease progression as by RECIST v1.1 per Investigator's Review or death due to any cause, whichever occurred first. Objective progression was defined as a 20% increase in the sum of the diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm or unequivocal progression of pre-existing non-target lesions, or the appearance of any new unequivocal malignant lesions. Tumor tissue from participants' original diagnostic biopsies or recently obtained biopsies were analyzed to determine KRAS status.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 256 | 263
Months | 1.9 [1.8 to 2.7] | 1.9 [1.8 to 2.6]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Test type: Superiority or Other; p = 0.728, 1-sided stratified log-rank test — One-sided P-value; Stratified by EGFR status and baseline ECOG; Hazard Ratio (HR) = 1.057, 95% CI 2-sided [0.881 to 1.267] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Overall Survival (OS).
Description: OS was defined as the time from randomization to the date of death for any cause. In the absence of confirmation of death, survival time was censored at the last date the patient was known to be alive (ie, at their last known alive date from long term follow-up).
Time Frame: From date of randomization until the date of death from any cause or last date known to be alive, participants were followed up regardless of the reason for discontinuation from study treatment at intervals of no longer than every 2 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 439 | 439
Months | 7.9 [6.8 to 9.0] | 8.3 [7.4 to 9.7]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Test type: Superiority or Other; p = 0.638, 1-sided stratified log-rank test. — One-sided P-value; Stratified by EGFR status, KRAS status, and baseline ECOG; Hazard Ratio (HR) = 1.026, 95% CI 2-sided [0.887 to 1.188] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: OS in KRAS-WT Participants.
Description: OS was defined as the time from randomization to the date of death for any cause. In the absence of confirmation of death, survival time was censored at the last date the patient was known to be alive (ie, at their last known alive date from long term follow-up). Tumor tissue from participants' original diagnostic biopsies or recently obtained biopsies were analyzed to determine KRAS status.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 256 | 263
Months | 8.1 [6.7 to 9.4] | 8.5 [7.5 to 10.2]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Test type: Superiority or Other; p = 0.775, 1-sided stratified log-rank test. — One-sided P-value; Stratified by EGFR status and baseline ECOG; Hazard Ratio (HR) = 1.078, 95% CI 2-sided [0.886 to 1.312] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Best Overall Response (BOR) Per Independent Radiologic Review.
Description: The BOR was the best response per RECIST (version 1.1) criteria as assessed by independent assessment recorded from randomization until disease progression. Per RECIST version 1.1: Complete Response (CR): disappearance of all pre-existing lesions except nodal disease, with all nodal lesions decreased to normal size (short axis<10 mm) and no appearance of new unequivocal malignant lesions; Partial Response (PR): >=30% decrease from baseline sum of diameters of all target lesions with no unequivocal progression of pre-existing non-target lesions or appearance of new unequivocal malignant lesions; Progressive Disease (PD): >=20% increase in the sum of diameters of target lesions above the smallest sum observed, with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions.
Time Frame: From date of randomization until progression or initiation of new anti-cancer therapy or death. Participants were followed up until progressive disease regardless of start of subsequent cancer therapy.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 439 | 439
Participants
  Complete response | 6 | 8
  Partial response | 46 | 27
  Stable/No response | 163 | 182
  Objective progression | 151 | 146
  Indeterminate | 73 | 76

8. Secondary Outcome: BOR Per Investigator Review.
Description: The BOR was the best response per RECIST (version 1.1) criteria as assessed by investigator assessment recorded from randomization until disease progression. Per RECIST version 1.1: CR: disappearance of all pre-existing lesions except nodal disease, with all nodal lesions decreased to normal size (short axis<10 mm) and no appearance of new unequivocal malignant lesions; PR: >=30% decrease from baseline sum of diameters of all target lesions with no unequivocal progression of pre-existing non-target lesions or appearance of new unequivocal malignant lesions; PD: >=20% increase in the sum of diameters of target lesions above the smallest sum observed, with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 439 | 439
Participants
  Complete response | 2 | 3
  Partial response | 57 | 42
  Stable/No response | 136 | 136
  Objective progression | 191 | 206
  Indeterminate | 53 | 52

9. Secondary Outcome: Duration of Response (DR) Based on Independent Radiologic Review.
Description: DR was defined as the time from first documentation of response assessed by independent review (CR or PR whichever occurred first) to date of progression or death due to any cause, whichever occurs first. Per RECIST version 1.1: CR: disappearance of all pre-existing lesions except nodal disease, with all nodal lesions decreased to normal size (short axis<10 mm) and no appearance of new unequivocal malignant lesions; PR: >=30% decrease from baseline sum of diameters of all target lesions with no unequivocal progression of pre-existing non-target lesions or appearance of new unequivocal malignant lesions; PD: >=20% increase in the sum of diameters of target lesions above the smallest sum observed, with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions.
Time Frame: From date of randomization until progression or death due to any cause. Participants were followed up until progressive disease regardless of start of subsequent cancer therapy.
Population: DR was analyzed for a subgroup of participants in the ITT population, who had an objective tumor response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 52 | 35
Months | 9.2 [6.9 to 20.2] | 10.1 [5.6 to 14.8]

10. Secondary Outcome: DR Based on Investigator Review.
Description: DR was defined as the time from first documentation of response assessed by investigator review (CR or PR whichever occurred first) to date of progression or death due to any cause, whichever occurs first. Per RECIST version 1.1: CR: disappearance of all pre-existing lesions except nodal disease, with all nodal lesions decreased to normal size (short axis<10 mm) and no appearance of new unequivocal malignant lesions; PR: >=30% decrease from baseline sum of diameters of all target lesions with no unequivocal progression of pre-existing non-target lesions or appearance of new unequivocal malignant lesions; PD: >=20% increase in the sum of diameters of target lesions above the smallest sum observed, with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions or appearance of any new unequivocal malignant lesions.
Time Frame: as for outcome 9
Population: DR was analyzed for a subgroup of participants in the ITT population, who had an objective tumor response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 59 | 45
Months | 10.4 [7.4 to 16.6] | 9.2 [6.2 to 11.3]

11. Secondary Outcome: Trough Concentrations (Ctrough) of Dacomitinib.
Description: Mean Ctrough values of dacomitinib observed from Cycle 2 through 5, Day 1 for dose compliant participants.
Time Frame: Baseline up to Cycle 5 Day 1
Population: Participants treated with dacomitinib with at least one measured plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Trough Plasma Concentration (ng/mL)
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo)
Number analyzed (Participants) | 317
Trough Plasma Concentration (ng/mL)
  Cycle (C) 2 Day (D) 1 (n=317) | 61.0102 (77)
  C3D1 (n=175) | 46.5229 (97)
  C4D1 (n=131) | 44.2708 (86)
  C5D1 (n=95) | 38.0307 (83)

12. Secondary Outcome: Trough Concentrations (Ctrough) of PF-05199265.
Description: Mean Ctrough values of PF-05199265 observed from Cycle 2 through 5, Day 1 for dose compliant participants.
Time Frame: Baseline up to Cycle 5 Day 1
Population: Participants treated with dacomitinib with at least one measured plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Trough Plasma Concentration (ng/mL)
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo)
Number analyzed (Participants) | 323
Trough Plasma Concentration (ng/mL)
  Cycle (C) 2 Day (D) 1 (n=323) | 6.3695 (129)
  C3D1 (n=179) | 5.8706 (123)
  C4D1 (n=136) | 6.4380 (116)
  C5D1 (n=100) | 6.5353 (118)

13. Secondary Outcome: Time to Deterioration (TTD) in Pain, Dyspnea, Fatigue or Cough Patient Reported Disease Symptoms.
Description: TTD defined as the time from first dose (baseline) to the first time a patient's score in pain, dyspnea, fatigue or cough from the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (QLQ-LC13) increased by ≥10 points. A ≥10 point increase in score had to be maintained for ≥2 consecutive cycles for the symptom to be considered deteriorated. Participants were censored at the last time when they completed an assessment for pain, dyspnea, fatigue or cough if they had not deteriorated. A 10 point or higher change in the score is perceived by participants as clinically significant.
Time Frame: Data taken from Cycle 1 day 1 to the end of treatment or withdrawal.
Population: The PRO analysis set included all participants who started treatment and completed the baseline and at least 1 post-dosing PRO assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 421 | 424
Months | 1.0 [1.0 to 1.9] | 1.0 [0.9 to 1.4]

14. Secondary Outcome: Mean and Difference in Mean in Functioning and Global Quality of Life (QOL) as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Scores ranged from 0-100 where a higher score indicated a better level of quality of life. Overall scores present the mean score for that scale from all time-point data.
Time Frame: Data taken from Cycle 1 day 1 to the end of treatment or withdrawal, averaged (mean) to provide overall scores.
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Units on a scale.
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 421 | 424
Units on a scale.
  QLQ-C30 Global QoL | 56.4068 [54.631 to 58.183] | 58.3425 [56.554 to 60.131]
  QLQ-C30 Cognitive Functioning | 83.8980 [82.275 to 85.521] | 83.0913 [81.461 to 84.722]
  QLQ-C30 Emotional Functioning | 79.1982 [77.390 to 81.007] | 78.4682 [76.658 to 80.279]
  QLQ-C30 Physical Functioning | 75.2138 [73.250 to 77.210] | 73.6849 [71.719 to 75.651]
  QLQ-C30 Role Functioning | 69.3252 [66.771 to 71.879] | 68.1033 [65.553 to 70.653]
  QLQ-C30 Social Functioning | 74.7868 [72.371 to 77.203] | 76.2839 [73.864 to 78.703]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Global QoL. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.9357, 95% CI [-4.278 to 0.407] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 2: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 cognitive functioning. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 0.8067, 95% CI [-1.312 to 2.926] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 3: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 emotional functioning. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model = 0.7300, 95% CI [-1.575 to 3.035] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 4: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 physical functioning. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 1.5289, 95% CI [-0.756 to 3.814] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 5: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 role functioning. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 1.2219, 95% CI [-1.975 to 4.419] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 6: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 social functioning. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.4970, 95% CI [-4.575 to 1.581] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)

15. Secondary Outcome: Mean and Difference in Mean in QLQ-C30 Symptoms as Assessed by the EORTC-QLQ-C30.
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Scores ranged from 0-100 where a higher score indicated a greater degree of symptoms/problems. Overall scores present the mean score for that scale from all time-point data.
Time Frame: Data taken from Cycle 1 day 1 to the end of treatment or withdrawal, averaged (mean) to provide overall scores.
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Units on a scale.
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 421 | 424
Units on a scale.
  QLQ-C30 Appetite loss | 28.5960 [25.841 to 31.351] | 27.3109 [24.532 to 30.090]
  QLQ-C30 Constipation | 8.2496 [6.392 to 10.108] | 14.1726 [12.299 to 16.046]
  QLQ-C30 Diarrhea | 38.8641 [36.303 to 41.425] | 18.6077 [16.017 to 21.198]
  QLQ-C30 Dysponea | 28.3313 [25.736 to 30.927] | 32.8812 [30.282 to 35.480]
  QLQ-C30 Fatigue | 35.0885 [32.848 to 37.329] | 36.7469 [34.494 to 38.999]
  QLQ-C30 Financial Difficulties | 20.0597 [17.760 to 22.360] | 20.0597 [17.760 to 22.360]
  QLQ-C30 Insomnia | 19.7903 [17.413 to 22.168] | 24.6615 [22.276 to 27.046]
  QLQ-C30 Nausea and Vomiting | 9.1438 [7.759 to 10.528] | 9.6362 [8.208 to 11.065]
  QLQ-C30 Pain | 25.1850 [22.867 to 27.503] | 24.8754 [22.551 to 27.200]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Appetite loss. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 1.2851, 95% CI 2-sided [-2.416 to 4.986] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 2: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Constipation. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -5.9230, 95% CI 2-sided [-8.432 to -3.414] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 3: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Diarrhea. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model = 20.2564, 95% CI 2-sided [16.874 to 23.639] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 4: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Dysponea. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -4.5499, 95% CI 2-sided [-7.719 to -1.381] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 5: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Fatigue. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.6584, 95% CI 2-sided [-4.442 to 1.125] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 6: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Financial Difficulties. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -0.1469, 95% CI [-3.056 to 2.762] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 7: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Insomnia. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -4.8711, 95% CI 2-sided [-7.998 to -1.745] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 8: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Nausea and Vomiting. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -0.4924, 95% CI 2-sided [-2.485 to 1.500] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 9: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for QLQ-C30 Pain. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 0.3096, 95% CI 2-sided [-2.646 to 3.265] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)

16. Secondary Outcome: Mean and Difference in Mean in Lung Cancer Symptom Scores as Assessed by the EORTC QLQ- LC13.
Description: The QLQ-LC13 included questions specific to the disease associated symptoms (dyspnea, cough, haemoptysis, and site specific pain), treatment-related symptoms (sore mouth, dysphagia, neuropathy, and alopecia), and analgesic use of lung cancer patients. Scores range from 0-100 and a higher score indicates greater degree of symptoms/problems. Overall scores present the mean score for that scale from all time-point data.
Time Frame: Data taken from Cycle 1 day 1 to the end of treatment or withdrawal, averaged (mean) to provide overall scores.
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Units on a scale.
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 421 | 424
Units on a scale.
  QLQ-LC13 Trouble Swallowing | 10.1934 [8.360 to 12.027] | 7.5553 [5.711 to 9.400]
  QLQ-LC13 Coughing | 28.3790 [26.037 to 30.721] | 32.6294 [30.272 to 34.986]
  QLQ-LC13 Haemoptysis | 3.4751 [2.118 to 4.832] | 4.5515 [2.615 to 6.488]
  QLQ-LC13 Sore Mouth | 20.4054 [18.115 to 22.696] | 11.0509 [8.731 to 13.371]
  QLQ-LC13 Shortness of Breath | 27.1651 [25.161 to 29.169] | 28.3413 [26.346 to 30.337]
  QLQ-LC13 Peripheral Neuropathy | 19.4905 [17.222 to 21.759] | 20.1284 [17.850 to 22.407]
  QLQ-LC13 Alopecia | 14.8327 [11.848 to 17.818] | 16.1963 [13.220 to 19.173]
  QLQ-LC13 Pain in Chest | 16.4268 [14.335 to 18.518] | 17.6430 [15.541 to 19.745]
  QLQ-LC13 Pain in Arm or Shoulder | 15.9840 [13.864 to 18.104] | 17.1315 [14.989 to 19.274]
  QLQ-LC13 Pain in other Parts | 21.5437 [19.020 to 24.067] | 22.6124 [20.060 to 25.165]
  QLQ-LC13 Any Med for Pain | 61.8437 [58.169 to 65.519] | 61.8115 [58.038 to 65.585]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Trouble Swallowing as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 2.6381, 95% CI [0.172 to 5.104] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 2: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Coughing as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -4.2504, 95% CI [-7.178 to -1.322] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 3: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Haemoptysis as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model = -1.0764, 95% CI [-3.997 to 1.845] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 4: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Sore Mouth as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 9.3545, 95% CI [6.211 to 12.497] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 5: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Shortness of Breath as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.1762, 95% CI [-3.560 to 1.208] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 6: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Peripheral Neuropathy as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -0.6378, 95% CI [-3.684 to 2.408] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 7: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Alopecia as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.3637, 95% CI [-4.546 to 1.819] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 8: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Pain in Chest as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.2163, 95% CI [-3.885 to 1.452] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 9: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Pain in Arm or Shoulder as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.1475, 95% CI [-3.902 to 1.607] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 10: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Pain Other Parts as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -1.0687, 95% CI [-4.488 to 2.351] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)
Statistical Analysis 11: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for Any Med for Pain as Assessed by the EORTC-QLQ-LC13. Estimated change from baseline was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-LC13 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = 0.0322, 95% CI [-4.847 to 4.911] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)

17. Secondary Outcome: Mean and Difference in Mean of the EuroQoL-5 Dimensions (EQ-5D) Visual Analogue Scale (VAS) Score
Description: The EQ-5D is a validated and reliable self-report preference-based measure developed by the EuroQoL Group to assess health-related quality of life. It consists of the EQ-5D descriptive system and a visual analogue scale-the EQ VAS. The EQ-5D descriptive system measures a participants' health state on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels, reflecting "no health problems," "moderate health problems," and "extreme health problems." The EQ VAS records the respondent's self-rated health on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Data taken from Cycle 1 day 1 to the end of treatment or withdrawal, averaged (mean) to provide overall scores.
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: Units on a scale.
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Number analyzed (Participants) | 421 | 424
Units on a scale. | 65.1908 [63.519 to 66.863] | 65.5794 [63.908 to 67.250]
Statistical Analysis 1: Comparison: Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) vs Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo); Analysis presented for EQ-5D VAS. Mean difference was from a repeated measures mixed-effects model with an intercept term, treatment, treatment-by-time interaction, and baseline EORTC QLQ-C30 subscale baseline score (intercept and time from first dose are included as random effects). Confidence intervals provided were not adjusted for multiplicity; Test type: Superiority or Other; Repeated measures mixed-effects model. = -0.3886, 95% CI [-2.413 to 1.636] — This analysis represents the mean difference between the dacomitinib arm (Arm A) and the erlotinib arm (Arm B)

ADVERSE EVENTS:
Time Frame: AE reporting period is from 1st dose of study drug through 28 days after last dose of study drug. SAE reporting period is from informed consent through 28 days after last dose of study drug. The longest duration of treatment in this study was 48 weeks.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo)
Serious Adverse Events (participants affected / at risk) | 178/436 | 169/436
Other Adverse Events (participants affected / at risk) | 424/436 | 417/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) (N=436) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo) (N=436)
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 3
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 20 | 7
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3
Asthenia (General disorders) | 3 | 2
Axillary pain (General disorders) | 0 | 1
Catheter site pain (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 2
Condition aggravated (General disorders) | 3 | 2
Death (General disorders) | 5 | 1
Disease progression (General disorders) | 53 | 48
Drug interaction (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 4
General physical health deterioration (General disorders) | 4 | 10
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 0
Pain (General disorders) | 0 | 2
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Acne pustular (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 12 | 15
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 3
Rhinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 3
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Aspiration bronchial (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 13 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 2
Renal impairment (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Internal fixation of fracture (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Embolism (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Blinded Dacomitinib and Blinded Erlotinib Placebo) (N=436) | Arm B (Blinded Erlotinib and Blinded Dacomitinib Placebo) (N=436)
Anaemia (Blood and lymphatic system disorders) | 35 | 43
Tachycardia (Cardiac disorders) | 5 | 10
Dry eye (Eye disorders) | 16 | 5
Abdominal pain (Gastrointestinal disorders) | 21 | 19
Abdominal pain upper (Gastrointestinal disorders) | 21 | 20
Cheilitis (Gastrointestinal disorders) | 13 | 8
Constipation (Gastrointestinal disorders) | 43 | 59
Diarrhoea (Gastrointestinal disorders) | 322 | 217
Dry mouth (Gastrointestinal disorders) | 14 | 13
Dyspepsia (Gastrointestinal disorders) | 20 | 16
Dysphagia (Gastrointestinal disorders) | 16 | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 11
Nausea (Gastrointestinal disorders) | 90 | 81
Stomatitis (Gastrointestinal disorders) | 81 | 52
Vomiting (Gastrointestinal disorders) | 71 | 70
Asthenia (General disorders) | 65 | 59
Chest pain (General disorders) | 21 | 36
Fatigue (General disorders) | 78 | 92
General physical health deterioration (General disorders) | 9 | 11
Malaise (General disorders) | 9 | 7
Mucosal inflammation (General disorders) | 67 | 28
Oedema peripheral (General disorders) | 17 | 29
Pain (General disorders) | 12 | 21
Pyrexia (General disorders) | 41 | 36
Xerosis (General disorders) | 14 | 7
Conjunctivitis (Infections and infestations) | 29 | 14
Cystitis (Infections and infestations) | 9 | 5
Lower respiratory tract infection (Infections and infestations) | 5 | 9
Nasopharyngitis (Infections and infestations) | 19 | 20
Paronychia (Infections and infestations) | 94 | 44
Rash pustular (Infections and infestations) | 9 | 9
Respiratory tract infection (Infections and infestations) | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 13 | 12
Urinary tract infection (Infections and infestations) | 18 | 19
Fall (Injury, poisoning and procedural complications) | 8 | 10
Alanine aminotransferase increased (Investigations) | 8 | 22
Aspartate aminotransferase increased (Investigations) | 10 | 21
Blood bilirubin increased (Investigations) | 0 | 11
Blood creatinine increased (Investigations) | 17 | 13
Weight decreased (Investigations) | 64 | 38
Decreased appetite (Metabolism and nutrition disorders) | 138 | 119
Dehydration (Metabolism and nutrition disorders) | 26 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 30
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 26
Dizziness (Nervous system disorders) | 17 | 25
Dysgeusia (Nervous system disorders) | 34 | 22
Headache (Nervous system disorders) | 18 | 20
Anxiety (Psychiatric disorders) | 16 | 19
Depression (Psychiatric disorders) | 7 | 9
Insomnia (Psychiatric disorders) | 14 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 54 | 73
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 76 | 81
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37 | 23
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 23 | 37
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Acne (Skin and subcutaneous tissue disorders) | 23 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 18
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 81 | 88
Dry skin (Skin and subcutaneous tissue disorders) | 86 | 84
Erythema (Skin and subcutaneous tissue disorders) | 18 | 21
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 49 | 54
Rash (Skin and subcutaneous tissue disorders) | 218 | 203
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 12
Skin exfoliation (Skin and subcutaneous tissue disorders) | 15 | 10
Skin fissures (Skin and subcutaneous tissue disorders) | 24 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No